CLINICAL TRIAL: NCT05441462
Title: Defining in Vivo Kinematics of Single Piece Silastic Joint Replacements in the Hand With Magnetic Resonance Imaging
Brief Title: Kinematics of Silastic Joint Replacements in the Hand
Status: Completed | Type: Observational
Sponsor: Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PIPJ
Record Dates: First submitted 2022-05-03; First posted 2022-07-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Degenerative Arthritis; Inflammatory Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Silastic Joint Replacement — Participants who have had silastic joint replacement surgery for degenerative or inflammatory arthritis within the last three years

SUMMARY:
To assess in vivo the kinematics of single piece silastic joint replacements in the hand with magnetic resonance imaging

DETAILED DESCRIPTION:
Proximal inter phalangeal joint (PIPJ) replacement is performed for pain relief in the end stage of arthritis. Rheumatoid arthritis is the commonest indication in the metacarpophalangeal joint (MCPJ). In the PIPJ there is a more even spilt between degenerative and rheumatoid arthritis.

There are several options for PIPJ replacement currently licensed for use in the United Kingdom although data is not entered in to the National Joint Registry so the exact numbers and failure rates are unknown. Data from the Norwegian joint registry indicates that 99% of implanted MCPJ and PIPJ replacements are single piece silastic implants.

Three main prostheses represent the majority of implants used in the United Kingdom, Swanson, Sutter and Neuflex. All these implants have been shown in the literature to fracture either at the hinge or the distal stem - hinge interface. This is true of explants and in vitro simulator testing.

Long term survivorship in MCPJ and PIPJ replacement is below that of hip and knee replacement. One of the largest single series shows 63% survivorship at 17 year follow up but with radiological evidence of failure in at least two thirds. This compares poorly to the 82.9% survivorship for Exeter cemented hip replacements at 22 years. The long term aim of this project is to understand how the implants move. This will help explain failure in particular the newly observe hinge failure in Neuflex implants and provide ideas to improve these implants. Any modifications can be tested on the in vitro finger joint testing rig The method of MRI acquisition will be similar to that described in. This will require optimising. In order to limit movement to a sagittal displacement, a thermoplastic splint will support the wrist and hand up to the level of the proximal palmer crease. A rig will also be made to hold the MCP / PIP joints in extension and positions of flexion increasing by 200 to maximum flexion. These will depend upon the patient's range of motion. The Investigators will define the centre of rotation of the hinge then points on the shoulder and stem of the implant from which to measure displacement. Points on the metacarpal and proximal phalanx will also be defined to allow measurement of the displacement of the implant relative to the bone during the range of movement.

ELIGIBILITY:
Inclusion Criteria:

- Single piece silastic joint replacement with an adequate range of movement (ROM), i.e.

an arc of movement of ≥ 50

* Age over 18
* Able to give informed consent

Exclusion Criteria:

* Any contraindication to MRI scanning
* Fractured implant
* Fixed flexion deformity >30 degrees in the replaced joint
* Total range of motion <50 degrees in the replaced joint
* Awaiting further surgery
* Abnormal joint instability
* Previous surgery on the same digit (other than the joint replacement)
* Replacement of the joint of the opposite hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are over the age of 18, able to give informed consent and have had a sialastic joint replacement and a native joint on the contralateral hand will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Deformation Assesment - Assesment of deformation of single piece silastic joint replacements in vivo | Six months
  Currently the only studies of single piece silastic joint replacement movements are in cadaveric models. These have shown there is a difference in the instantaneous centre of rotation between replacement and native joints. This has not been shown in vivo. As stated in the rational of the study the issue to address is the high failure rate of single piece silastic joint replacements in the hand. Key to this is understanding how they behave in vivo and how this differs from native joints. The primary objective is to show that in vivo displacement can be shown with MRI and is a reproducible method. Once the MRI scans have been obtained a computer generated 3D model of the scans will be made and measurements of deformation of the implant and its movements relative to the bony supporting structure will be made.

SECONDARY OUTCOMES:
To compare the movement of different implant designs and single replacements with native joints in combination with the assesment of acceptability and feasibility of MRI. | Through study completion, an average of one year
  As this is an observational study there is no endpoint set other than the completed acquisition of the MRI sequences and the measurement of PROMS for each patient in the form of the patient rated wrist evaluation score and the quick disability of arm, shoulder and hand score.

CONTACTS AND LOCATIONS:
Locations (1):
- Wrightington, Wigan & Leigh Teaching Hospitals NHS Foundation Trust, Wigan, United Kingdom

IPD SHARING:
Plan to Share IPD: No